CLINICAL TRIAL: NCT04820595
Title: Postoperative Neurocognitive Dysfunction: Is There Any Place for Emergency Agitation: A Prospective Cohort Trial
Acronym: PoD
Status: Completed | Type: Observational
Sponsor: Negovsky Reanimatology Research Institute (Other Government)
Responsible Party: Principal Investigator, Valery Likhvantsev, MD, Head of the Research Negovsky Reanimatology Research Institute, Negovsky Reanimatology Research Institute
Other Study IDs: PoD-2021
Record Dates: First submitted 2021-03-23; First posted 2021-03-29 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Emergence Delirium; Emergence Agitation; Postoperative Delirium
Keywords: emergence agitation; postoperative agitation; postoperative delirium; postoperative cognitive dysfunction; emergence delirium
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Patients who have RASS < +2 and have not delirium according CAM-ICU immediately upon emergence from anesthesia
  Interventions: Diagnostic Test: RASS; Diagnostic Test: CAM-ICU
- Agitated non-delirious group: Patients who have RASS = +2 or more and have not delirium according CAM-ICU immediately upon emergence from anesthesia
  Interventions: Diagnostic Test: RASS; Diagnostic Test: CAM-ICU
- Agitated delirium group: Patients who have RASS = +2 or more and have delirium according CAM-ICU immediately upon emergence from anesthesia
  Interventions: Diagnostic Test: RASS; Diagnostic Test: CAM-ICU

INTERVENTIONS:
Diagnostic Test: RASS — Richmond Agitation-Sedation Scale
Diagnostic Test: CAM-ICU — Confusion Assessment Method for the ICU

SUMMARY:
Perioperative neurocognitive disorders (PND) have been studying by clinicians, particularly by anesthesiologists, pretty long, however the most inspiring advancements were achieved during the last few decades. The most recent classification of PND which includes cognitive decline diagnosed before operation (described as neurocognitive disorder); any form of acute event (postoperative delirium) and cognitive decline diagnosed up to 30 days after the procedure (delayed neurocognitive recovery) and up to 12 months (postoperative neurocognitive disorder) was proposed in 2017. However at will one can notice at least one uncertainty that pertinent to the definition of delirium, emergency delirium and not mentioned in the classification discussed agitation.

The objective of the study is to determine if there is a difference between emergence agitation and emergence delirium.

ELIGIBILITY:
Inclusion Criteria:

* Age from 45 to 74 years
* Undergoing elective orthopedic surgery
* Provide written informed consent to participate in the PoD trial

Exclusion Criteria:

* Undergoing emergent/urgent surgery
* Montreal Cognitive Assessment < 18 points
* History of mental disorders according ICD-11
* Treated with at least one psychotropic drug
* Patients with neuromuscular disease
* Inability to undergo preoperative assessment for any reason
* Previously enrolled in PoD trial

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from 45 to 74 years old undergoing elective orthopedic surgery
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
frequency of postoperative delirium | 5 postoperative day
  Percent of postoperative delirium
frequency of postoperative cognitive dysfunction | 7 postoperative day
  Percent of postoperative cognitive dysfunction

SECONDARY OUTCOMES:
frequency of emergence agitation | immediately upon emergence from anesthesia
  Percent of emergence agitation
frequency of emergence delirium | immediately upon emergence from anesthesia
  Percent of emergence delirium
Length of postoperative delirium | 5 postoperative day
  Day of the end of postoperative delirium - day of onset of postoperative delirium
Length of stay in ICU | 1 year
  From ICU admission to ICU discharge
Length of hospitalization | 1 year
  From operative day to hospital discharge
MACE | 30 day
  Cardiac death or Myocardial infarction or Non-fatal cardiac arrest or Coronary revascularization
MACE | 1 year
  Cardiac death or Myocardial infarction or Non-fatal cardiac arrest or Coronary revascularization
MACCE | 30 day
  Cardiac death or Myocardial infarction or Non-fatal cardiac arrest or Coronary revascularization or Cerebrovascular accident
MACCE | 1 year
  Cardiac death or Myocardial infarction or Non-fatal cardiac arrest or Coronary revascularization or Cerebrovascular accident
30-day mortality | 30 day
  30-day mortality
1-year mortality | 1 year
  1-year mortality

CONTACTS AND LOCATIONS:
Overall Officials: Valery Likhvantsev, Principal Investigator — Negovsky Reanimatology Research Institute
Locations (2):
- Russia (2):
  - Moscow Scientific Clinical Center, Moscow
  - Main Military Clinical Hospital n.a. Acad.N. N. Burdenko, Moscow